CLINICAL TRIAL: NCT00659243
Title: A Prospective, Randomized, Double-blind Crossover Study Comparing 0.15 g/L rhBSSL Added to Pasteurized Breast Milk Versus Placebo During One Week of Treatment in Preterm Infants Born Before Week 32 of Gestational Age
Brief Title: Efficacy and Safety of Bile Salt Stimulated Lipase (BSSL) as Replacement Therapy in Pasteurized Breast Milk for Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BVT.BSSL-021
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Replacement Therapy in Preterm Infants
Keywords: Replacement therapy; Pasteurized breast milk; Preterm infants; BSSL

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhBSSL (Experimental)
  Interventions: Drug: rhBSSL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhBSSL — 0.15 g/L rhBSSL added to pasteurized breast milk; one week treatment
  Other Names: bucelipase alfa (INN)
  Arms: rhBSSL
Drug: Placebo — One week treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy in preterm infants following treatment with BSSL when administered in pasteurized breast milk.

DETAILED DESCRIPTION:
In this double-blind crossover study, patients will be randomized to receive pasteurized breast milk including BSSL or pasteurized breast milk without BSSL for the first 7 days. After a wash-out period of 2 days the patients will "crossover" to the other treatment regimen and receive an additional 7 days treatment. The primary efficacy measurements will be made by collecting stool during the last three days of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants
* less than or equal to 32 weeks of gestational age
* appropriate for gestational age
* enterally fed with pasteurized breast milk

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Coefficient of Fat Absorption measured in stool | Stool collected for a 72-hour period during the final 3 days of each treatment period

SECONDARY OUTCOMES:
Change in length and body weight | Baseline and after one week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Timdahl, MD, Study Director — Biovitrum AB
Locations (8):
- France (6):
  - Hopital de la Croix Rousse, Lyon
  - Hopital la Conception,, Marseille
  - Maternité A. Pinard, Néonatologie, Nancy
  - Hopital Saint Vincent de Paul, Paris
  - Hopital des Enfants, Toulouse
  - CHRU de Tours, Centre de Pédiatrie Gatien de Clocheville, Tours
- Italy (2):
  - Presidio Ospedaliero di Alta Specializzazione G.Salesi Azienda Ospedaliero Universitaria Ospedali Riuniti "Umberto I-G.M. Lancisi-G.Salesi", Ancona
  - Policlinico Universitario-Azienda Ospedeliero di Padova, Dipartimento di Pediatria, Padua

REFERENCES:
- [Derived] Casper C, Carnielli VP, Hascoet JM, Lapillonne A, Maggio L, Timdahl K, Olsson B, Vagero M, Hernell O. rhBSSL improves growth and LCPUFA absorption in preterm infants fed formula or pasteurized breast milk. J Pediatr Gastroenterol Nutr. 2014 Jul;59(1):61-9. doi: 10.1097/MPG.0000000000000365. PMID 25222806